CLINICAL TRIAL: NCT03841461
Title: Investigation of the Effect of Physical Activity Level on Sleep Quality and Fatigue in Academicians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 284
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Physical Activity; Sleep; Fatigue
Keywords: Academician; Physical Activity Level; Sleep Quality; Fatigue
MeSH Terms: conditions — Motor Activity; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Academicians: The academicians working in any program of any higher education institution
  Interventions: Other: International Physical Activity Questionnaire-Short Form; Other: The Pittsburgh Sleep Quality Index; Other: The Fatigue Severity Scale; Other: General Information Form

INTERVENTIONS:
Other: International Physical Activity Questionnaire-Short Form — IPAQ has been developed to obtain valid and comparable information about the level of physical activity based on individual reports on daily physical activity in the international arena. This form consists of 7 questions; provides information about time spent in walking, moderate and violent activities, and time spent sitting. The calculation of the total score of the short form includes total of duration and frequency whom walking, moderate activity and severe activity. The energy required for the activities is calculated by the MET-minute score.Standard MET values for these activities has been established. These; Walking = 3.3 MET;Moderate Severe Physical Activity = 4.0 MET;Severe Physical Activity = 8.0 MET;Seating = 1.5 MET.Classification is based on the numerical data obtained.Accordingly,there are 3 activity levels: Inactive,minimal active and very active.
  Other Names: IPAQ-SF
Other: The Pittsburgh Sleep Quality Index — It is a scale that provides information about the sleep quality of the individuals and the type and severity of the sleep disorder in the last month. It consists of 24 questions, 19 of which are evaluated. The PSQI consists of 1 total score and 7 sub-dimensions (subjective sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disturbance, sleep medication use, daytime dysfunction). Each item in the scale has a value between 0 (no distress) and 3 (serious distress). The sum of the scores related to the seven sub-dimensions gives the total PSQI score. The score of each sub-dimension ranges from 0 to 3. The total PSQI score ranged from 0 to 21. While the sleep quality of the patients with a total score of 5 and below is considered as 'good'; >5 refers to poor sleep quality.
  Other Names: PSQI
Other: The Fatigue Severity Scale — Each question on this scale, which is composed of Likert type questions: 1.I strongly disagree 2.I do not agree 3.No tend to disagree 4. Indefinitely. The score of the scale, which consists of 9 questions, varies between 9-63. People are asked to mark the appropriate options for each question taking into account their status in the last 1 month period.
  Other Names: FSS
Other: General Information Form — A form, which is prepared by us, including the purpose of the study, demographic information, daily working hours and assignment durations.

SUMMARY:
Physical activity is closely associated with well-being condition and health development. The sleep quality and fatigue levels of individuals are also important components of health. Within the scope of our study, it is aimed to investigate the physical activity levels, sleep quality and fatigue levels of the academicians, who are generally working on a desk and we think that they live a sedentary life. Within the scope of this study, academicians were asked to respond to , International Physical Activity Questionnaire-Short Form (IPAQ-Short Form), general evaluation form, Pittsburg Sleep Quality Index (PSQI) and Fatigue Severity Scale (FSS) .

DETAILED DESCRIPTION:
The aim of this study is to investigate that the effect of physical activity level on sleep quality and fatigue in academicians.

First of all, a form including the purpose of the study, demographic information, daily working hours and assignment durations, was arranged; then obtaining general information about academicians who participated in the study and the physical activity levels of the individuals with International Physical Activity Questionnaire-Short Form (IPAQ-Short Form); sleep quality with the Pittsburg Sleep Quality Index (PSQI); fatigue levels with Fatigue Severity Scale (FSS) were planned to be measured. On-line communication was preferred as a data collection tool for all these assessments. In order to prevent bias in the results of the study, it was planned to transmit the questionnaire on-line to the academicians working in any program of any higher education institution. In this way, the voluntary involvement of the participant or any other threat to abuse was prevented. In other words, it was planned to ensure that individuals answer or don't respond the form on a purely voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

Volunteering, to work as academicians in any department of any higher education institution.

Exclusion Criteria:

refuse to participate in the study, not being an academician

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The academicians working in any department of any higher education institution.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
The level of physical activity | 1 month
  International Physical Activity Questionnaire-Short Form (IPAQ-SF) consists of 7 questions;provides information about the level of physical activity in the last 7days.The calculation of the total score of the form includes total of duration and frequency whom walking,moderate activity and severe activity.The MET-minute scores;Walking 3.3MET,Moderate Severe Physical Activity 4MET,Severe Physical Activity 8MET,Seating 1.5MET.Classification is based on the numerical data obtained.Accordingly,there are 3 activity levels: Inactive,minimal active and very active.The lowest level of physical activity is inactive and the highest level of physical activity is very active.

SECONDARY OUTCOMES:
Sleep Quality | 1 month
  The Pittsburgh Sleep Quality Index (PSQI) is a scale that provides information about the sleep quality of the individuals and the type and severity of the sleep disorder in the last month. It consists of 24 questions, 19 of which are evaluated. The PSQI consists of 1 total score and 7 sub-dimensions (subjective sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disturbance, sleep medication use, daytime dysfunction). Each item in the scale has a value between 0 (no distress) and 3 (serious distress). The sum of the scores related to the seven sub-dimensions gives the total PSQI score. The score of each subdimension ranges from 0 to 3. The total PSQI score ranged from 0 to 21. While the sleep quality of the patients with a total score of 5 and below is considered as 'good'; >5 refers to poor sleep quality.
Fatigue Level | 1 month
  Fatigue Severity Scale (FSS) is one of the most commonly used self-report questionnaires to measure fatigue. Each question on this scale, which is composed of Likert type questions: 1.I strongly disagree 2.I do not agree 3.No tend to disagree 4. Indefinitely. The total score of the scale, which consists of 9 questions, varies between 9-63. People are asked to mark the appropriate options for each question taking into account their status in the last 1 month period. A total of 36 points and above indicate fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Nazire Nur Yıldız, PT, Principal Investigator — AYBU Institute of Health Sciences Department of Physiotherapy and Rehabilitation Master Program/Master Degree Student; Ertuğrul Demirdel, Asst. Prof., Principal Investigator — AYBU Faculty of Health Sciences Department of Physiotherapy and Rehabilitation
Locations (1):
- Ankara Yıldırım Beyazıt University, Institute of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Province, Turkey (Türkiye)